CLINICAL TRIAL: NCT03887741
Title: Plasmapheresis Versus Plasma Infusion from Young APOE3 Homozygotes Into MCI APOE4 Homozygotes to Slow Disease Progression: an Unblinded Phase 1 Safety, Methodological and Exploratory Biomarkers Study.
Brief Title: Plasmapheresis Versus Plasma Infusion from Young APOE3 Homozygotes Into MCI APOE4 Homozygotes to Slow Disease Progression
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Neill R. Graff-Radford, M.D., Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-007034
Record Dates: First submitted 2019-03-21; First posted 2019-03-25 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Plasmapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Plasmapheresis (Experimental): 3 patients will have monthly plasmapheresis for 6 months and followed for a total of 12 months
  Interventions: Biological: Plasmapheresis
- Plasma infusion (Experimental): 3 patients will have biweekly plasma infusion for 6 months and followed for 12 months
  Interventions: Biological: Plasma infusion
- Control group (No Intervention): 3 patients will be followed for 12 months

INTERVENTIONS:
Biological: Plasmapheresis — Patient will have monthly plasma exchange with young ApoE 33 plasma. Each exchange will be 1.5 volume of patient's plasma
  Arms: Plasmapheresis
Biological: Plasma infusion — Infuse every two weeks with ApoE33 young plasma (1unit) for 6 months
  Arms: Plasma infusion

SUMMARY:
Determine safety of plasma infusion or exchange in APOE 44 patients.

ELIGIBILITY:
Inclusion criteria

* Patient age 50 to 75.
* APOE 44 homozygote.
* Meets the Petersen criteria for MCI (41).
* Clinical Dementia Rating (CDR) of 0.5 and Mini Mental Status Examination (MMSE) of 24 to 30 inclusive.
* Has an informant who the investigator judges has sufficient patient contact to provide accurate information.
* Stable depression and or anxiety.
* Stable psychoactive medication for 6 weeks.

Exclusion criteria

* History of severe reaction to plasma or plasma derived products which include but not limited to severe allergic reaction, anaphylactic reaction and transfusion related acute lung injury (TRALI).
* Patients who do not want to receive blood transfusion for religious or cultural reasons such as Jehovah Witness Faith.
* Has a medical condition that would interfere with participation such as congestive heart failure (New York Heart Association Class III or IV), unstable angina, moderate to severe renal impairment, liver failure, and poorly controlled diabetes.
* History of autoimmune disease considered clinically significant or requiring chronic steroid or immune suppression medication.
* History of being HIV +.
* History of +VE test result indicating active hepatitis C or B (defined as both hepatitis B surface antigen and hepatitis core antibody +VE).
* Uncontrolled hypertension as defined by systolic/diastolic BP three times more than 165/100.
* No venous access for plasma exchange therapy.
* Any neurological condition that could be contributing to cognitive decline such as Lewy body disease, front temporal dementia, strokes or other cerebrovascular disease, head trauma, substance abuse, multiple sclerosis, Vitamin B12 deficiency, thyroid deficiency.
* Epileptic seizures within 10 years of screening.
* Cancer diagnosis (other than non-melanoma skin cancer) in the last 5 years.
* More than 1 subcortical stroke or more than 1 cortical stroke.
* Unable to have an MRI.
* MRI showing acute or subacute hemorrhage, evidence of normal pressure hydrocephalus, hemispheric infarcts, glioma or other brain tumor that could contribute to cognitive decline.
* Unstable psychiatric condition.
* On another experimental treatment study or has been on one in the last 3 months.
* If a patient consents to lumbar puncture (LP), they will be excluded from LP if any contraindication to having an LP is present. Examples are platelet count<100,000, spine deformity or contraindication to come off blood thinner for the LP. Patients may still participate in the rest of the study without having and LP.
* Any unspecified reason that the investigator finds the patient unsuitable to take part.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2024-02-16 (Actual); Study Completion 2024-02-16 (Actual)

PRIMARY OUTCOMES:
Adverse events | One year
  Number of adverse events reported

CONTACTS AND LOCATIONS:
Overall Officials: Neill R Graff-Radford, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials